CLINICAL TRIAL: NCT02804360
Title: Dexamethasone in Retinitis Pigmentosa Cystoid Macular Edema
Brief Title: Intravitreal Dexamethasone Implant in Retinitis Pigmentosa-related Macular Edema- a Retrospective Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rafic Hariri University Hospital (Other)
Responsible Party: Principal Investigator, Ahmad Mansour, MD, Clinical Professor, AUB, Chair, Department of Opthalmology, Rafic Hariri Hospital, Rafic Hariri University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INV-2016-267
Record Dates: First submitted 2016-05-18; First posted 2016-06-17 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Retinitis Pigmentosa; Cystoid Macular Edema
MeSH Terms: conditions — Retinitis Pigmentosa; Macular Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- therapy (Experimental): Dexamethasone injection
  Interventions: Device: dexamethasone injection

INTERVENTIONS:
Device: dexamethasone injection — intravitreal dexamethasone in retinitis pigmentosa cystoid macular edema
  Other Names: OZURDEX

SUMMARY:
Purpose: Cystoid macular edema (CME) in retinitis pigmentosa (RP) has been managed in several ways with little success. The aim of our study was to report the use of intravitreal dexamethasone implant in a large series of patients with RP and CME.

Setting: Retrospective case series. Methods: Cases were diagnosed as RP based on the classic fundus triad of bone-spicule pigment deposits (intraretinal pigmentary migration), retinal vessel attenuation, waxy pallor of the optic disc along with night blindness and attenuated ERG amplitudes (delays in rod or cone b-wave implicit times). Family history of RP and family screening for RP were important in establishing the diagnosis in eyes with some diagnostic challenge. CME was diagnosed by intravitreous fluorescein angiography IVFA and spectral domain optical coherence tomography (SD-OCT). BCVA was monitored using Snellen visual acuity chart and CME was monitored by SD-OCT on follow-up visits.

DETAILED DESCRIPTION:
Introduction Retinitis pigmentosa (RP) is a group of inherited progressive retinal degenerations characterized by photoreceptor dysfunction primarily affecting the rods, followed by cones with worldwide prevalence of approximately one in 3,000-4,000 for a total of 2 million affected individuals all over the world. After rods die, cone photoreceptors gradually die resulting in constriction of visual fields and eventual blindness in many patients. There is presently no cure for RP where photoreceptor apoptosis plays a key role, but considerable effort is devoted to the search of rescue strategies. This condition can lead to blindness in the advanced stages of disease, when it involves the central retina. Also macular abnormalities appear frequently in RP leading to visual decline. CME is prevalent in 20-70% of RP patients and several treatment options were reported with variable success rates and with many side-effects. Therapies have included oral or topical carbonic anhydrase inhibitors, intravitreal VEGF antagonists, and periocular or intravitreal corticosteroids. The dexamethasone implant has been recently approved for the treatment of maculopathies related to diabetic retinopathy or retinal vein occlusion or uveitis. The current study explores the role of such implant in CME from RP.

Methods The investigators conducted a retrospective noncomparative study of the use of intravitreal dexamethasone implant in eyes with CME from RP. The study adhered to the tenets of the declaration of Helsinki. All patients signed an informed consent after detailed review of the benefits and complications of current therapy.

RP is defined as the presence of the triad of bone-spicule pigment deposits, retinal vessel attenuation and waxy pallor of the optic disc. Family history of RP, family screening for RP, and ERG recordings were ancillary tests in atypical RP. CME is defined as the presence of cystoid changes in the macula seen on linear scans by spectral domain OCT regardless of presence of retinal thickening (Gorovoy). Primary outcomes were best-corrected visual acuity and central macular thickness. Study duration was January 2012?? to December 2015 with all participants signing a formal consent. Inclusion criteria included naïve or previously treated CME. Exclusion criteria included diabetes mellitus, vitreous hemorrhage, macular ischemia, macular scar from subretinal fibrosis, corneal scar, infectious conjunctivitis, prior cataract or vitreous surgery, and inability to commit for long-term follow-up. Primary outcome measures included best-corrected visual acuity (BCVA) assessed by Snellen charts and central macular thickness (CMT, mean thickness in the central 1000-μm diameter area) using spectral domain optical coherence tomography (OCT). Intravenous fluorescein angiography was done at the initial exam using standard protocol with visualization of the retinal midperiphery. Comprehensive ocular examination including applanation tonometry was performed at baseline, and usually at month 1, months 2 and months 3 and thereafter. Ozurdex® (Allergan, Inc., Irvine, CA, USA) is an intravitreal rod shaped implant containing 0.7 mg dexamethasone in the Novadur® poly (D,L-lactide-co-glycolide solid polymer sustained-release drug delivery system. The implant was injected under sterile conditions using povidone iodine 5%, sterile lid speculum and topical anesthesia. Only one patient who was 9-year old received sedative agents in order to achieve patient cooperation. The single-use applicator was injected into the midvitreous through a self-sealing scleral injection 3,5 mm posterior to the limbus at the superotemporal or inferotemporal area. Genetic testing was not carried in the current case series.

Statistical analyses were done using SPSS version 22 (IBM Corporation, Chicago, Illinois) and Wilcoxon-Signed Rank Test with significance set at p-value of 0.05.

ELIGIBILITY:
Inclusion Criteria: Retinitis pigmentosa with cystoid macular edema -

Exclusion Criteria: infection, inability to consent, cataract, glaucoma, end-stage retinitis pigmentosa

-

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
visual gain measured as Snellen visual acuity | 4 months
  logMAR improvement after ozurdex implant

SECONDARY OUTCOMES:
resolution of macular edema by OCT | 4 months
  OCT measurement of macular thickness

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Mansour, MD, Principal Investigator — RHUH

IPD SHARING:
Plan to Share IPD: Yes
we can share data through excel sheet